CLINICAL TRIAL: NCT05794789
Title: "We Are an Active Family": Promoting Child Physical Activity Through Social Identity Formation in the Family System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Collaborators: Diabetes Canada (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Professor, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 23-0022
Record Dates: First submitted 2023-03-02; First posted 2023-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity; Social Identity
Keywords: Moderate to vigorous physical activity (MVPA); Childhood obesity; Type 2 Diabetes; Identity formation
MeSH Terms: conditions — Motor Activity; Social Identification; Pediatric Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PA education and planning condition (No Intervention): This group will receive sessions and information-based booklet and series of worksheets that provide a tangible knowledge translation product for the family. The material will consist of Canada's PA guidelines recommending 60 minutes of MVPA a day and a breakdown of ways for the parent to help their child achieve this PA, outlining three main domains of parental support (encouragement, logistical support, and PA together). The material also contains information about the benefits of PA for the child and how to plan for family PA. The material specifically includes a brainstorming exercise for parents where they list physical activities they think their children have found fun in the past. The investigators will provide this material as prompts/suggestions. This list helps create the template for PA planning by contextualizing what the parents would like to do with their kids. An additional two sessions will include education and planning material related to family healthy eating.
- Identity formation condition (Experimental): This group will receive the same content as the education+planning comparison condition but with two additional coaching sessions. The session will include short overviews of the benefits of PA as a family, brainstorming how a family can each assist each other in PA, and an activity for developing a family PA action plan. Behavior change techniques that align with these approaches and are included in the coaching session include identity salience, identity similarity, as well as identity fit and contrast. This will be supplemented by an organization of fun family PA roles for all members (e.g., activity planner, goal setter, supporter, etc.) to instill involvement as well as items (creation of a family PA t-shirt, family PA photos and display, etc.) to instill distinctiveness, which is a central feature of a social identity.
  Interventions: Behavioral: Social Identity

INTERVENTIONS:
Behavioral: Social Identity — This group will receive the same content as the education+planning as well as two additional sessions. This includes short overviews of the benefits of PA as a family, brainstorming how a family can each assist each other in PA, and an activity for developing a family PA action plan. Behavior change techniques such as identity salience, identity similarity, and identity fit and contrast are included in the coaching session include. This will be supplemented by an organization of fun family PA roles for all members (e.g., activity planner, goal setter, supporter, etc.) to instill involvement as well as items (creation of a family PA t-shirt, family PA photos and display, etc.) to instill distinctiveness, which is a central feature of a social identity. Worksheets and discussion will be included. The second session will involve only the parent(s) to focus on parental support identity and the content is based on the behavior change principles of self-identity theory.
  Arms: Identity formation condition

SUMMARY:
The purpose of our study is to explore the effectiveness of physical activity (PA) identity formation in the family system as a promotor of long-term PA. The primary research question is:

Does a family identity formation condition (with education+planning) result in increased child moderate- to vigorous-intensity PA (MVPA) compared to a standard comparison education and planning condition at six months? Hypothesis: Child MVPA will be higher for the identity formation condition in comparison to the more standard PA education+planning condition at six months.

DETAILED DESCRIPTION:
The secondary research questions will include:

1. Does the identity formation condition improve child health-related fitness outcomes compared to the education and planning condition at six months? Hypothesis: Child health-related fitness will be higher for the identity formation condition in comparison to the education and planning condition.
2. Can group differences among behavioural, and health-related fitness outcomes be explained through a mediation model? Hypothesis: The covariance of the assigned conditions (identity formation, planning + education) on child MVPA will be explained by parental support, and through parental support identity (i.e., manipulation check). In turn, the covariance between support and health-related outcomes will be explained by MVPA among conditions. In the case of null outcomes for research question #1, the investigators will instead explore a prediction model of these variables rather than a mediation model.
3. Is there an intergenerational, seasonal, or sex difference across primary outcomes by assigned condition? Hypothesis: Parents in the identity formation condition will show higher physical activity via some activities being performed with their children (as part of social identity) in comparison to the other condition. No differences in child sex or season are hypothesized based on past research.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be at least one parent with at least one child between the ages of 6 and 12 years.
* Families (parents and/or guardians and children) residing in Greater Victoria, Nanaimo, Ladysmith, Duncan, Vancouver, Richmond, Surrey, Burnaby, British Columbia.
* Children that participate in <60 minutes/day of moderate to vigorous physical activity (MVPA)

Exclusion Criteria:

* If child is meeting the current physical activity guidelines >=60 minutes a day of moderate to vigorous physical activity per day.
* If participant does not pass Physical Activity Readiness Questionnaire (PARQ)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in children's moderate to vigorous physical activity to 6 months | Baseline, 6 weeks, 3 months, and 6 months
  Children's physical activity will be quantified by accelerometry. Children will wear an accelerometer for a minimum of 6 hours per day for 7 days at baseline, 6 weeks, 3 months, and 6 months.

SECONDARY OUTCOMES:
Parent-child intergenerational activity via seven-day accelerometry | Baseline - 6 months
  Accelerometer model has a Bluetooth proximity detection feature that can determine the presence (e.g., same room in a house, at the park together) or absence of close proximity between two accelerometers. The outcome variable will be average minutes per day parents and children were both engaging in physical activity at the same time while in close proximity.
Parent-child intergenerational activity measured via parent self-report | Baseline - 6 months
  For self-reported PA, the the Godin Leisure-Time Exercise Questionnaire will be used.
Body Composition - Weight | Baseline - 6 months
  Weight (kg)
Body Composition - Height | Baseline - 6 months
  Height (cm)
Body Composition - Waist Circumference | Baseline - 6 months
  Waist circumference (cm)
Body Composition - Percentage Body Fat | Baseline - 6 months
  Percentage body fat will be measured using a bioelectric impedance scale
Cardiovascular Fitness (ie: predicted maximal aerobic power) | Baseline - 6 months
  Will be assessed during a submaximal exercise test called the mCAFT Step Test
Musculoskeletal Fitness | Baseline - 6 months
  Measured using grip strength
Musculoskeletal Endurance | Baseline - 6 months
  Measured doing curl ups and push ups
Musculoskeletal Power | Baseline - 6 months
  Measured doing vertical jump test
Musculoskeletal Flexibility | Baseline - 6 months
  Measured doing sit and reach test
The Multi-Process Action Control (MPAC) Constructs - Instrumental Attitude | Baseline - 6 months
  Measured by standardized measurement scale - 1-7 Likert-type scale (strongly disagree to strongly agree)
The Multi-Process Action Control (MPAC) Constructs - Affective Judgements | Baseline - 6 months
  Measured by standardized measurement scale - 1-7 Likert-type scale (strongly disagree to strongly agree)
The Multi-Process Action Control (MPAC) Constructs - Perceived Capability | Baseline - 6 months
  Measured by standardized measurement scale - 1-7 Likert-type scale (strongly disagree to strongly agree)
The Multi-Process Action Control (MPAC) Constructs - Perceived Opportunity | Baseline - 6 months
  Measured by standardized measurement scale - 1-7 Likert-type scale (strongly disagree to strongly agree)
Social Identity | Baseline - 6 months
  Measured by standardized measurement scale - 1-7 Likert-type scale (strongly disagree to strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Rhodes, PhD, Principal Investigator — University of Victoria; Chris Blanshard, PhD, Study Chair — Dalhousie University; Valerie Carson, PhD, Study Chair — University of Alberta; Kurt Smith, PhD, Study Chair — University of Victoria; Mark Beauchamp, PhD, Study Chair — University of British Columbia; Shaelyn Strachan, PhD, Study Chair — University of Manitoba; Leigh Vanderloo, PhD, Study Chair — ParticipACTION
Locations (2):
- Canada (2):
  - Psychology of Exercise, Health, and Physical Activity (PEHPA) Laboratory, University of British Columbia, Vancouver, British Columbia
  - Behavioural Medicine Lab, University of Victoria, Victoria, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Streight E, Beauchamp MR, Smith KJ, Blanchard CM, Carson V, Strachan SM, Vanderloo LM, Courtnall S, Rhodes RE. "We are an active family": a randomized trial protocol to evaluate a family-system social identity intervention to promote child physical activity. BMC Public Health. 2024 Sep 27;24(1):2605. doi: 10.1186/s12889-024-20024-8. PMID 39333930